CLINICAL TRIAL: NCT02668393
Title: An Open Label Phase I of Oral Nintedanib Plus Weekly Docetaxel Therapy in Patients With Locally Advanced or Metastatic Lung Adenocarcinoma After Failure of Platinum -Based First Line Chemotherapy
Brief Title: Nintedanib and Weekly Docetaxel in Lung Adenocarcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1199.224; 2015-000317-52 (EudraCT Number)
Record Dates: First submitted 2016-01-27; First posted 2016-01-29 (Estimated); Results first posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; nintedanib

ARMS (4):
- Level 0 (Other): Nintedanib low dose with docetaxel
  Interventions: Drug: Docetaxel; Drug: Nintedanib
- Level 1 (Other): Nintedanib medium dose with docetaxel
  Interventions: Drug: Docetaxel; Drug: Nintedanib
- Level 2 (Other): Nintedanib high dose with docetaxel
  Interventions: Drug: Docetaxel; Drug: Nintedanib
- Level 3 (Other): Nintedanib continuous high dose with docetaxel
  Interventions: Drug: Docetaxel; Drug: Nintedanib

INTERVENTIONS:
Drug: Docetaxel
Drug: Nintedanib — Low Dose
  Arms: Level 0
Drug: Nintedanib — Medium dose
  Arms: Level 1
Drug: Nintedanib — High dose
  Arms: Level 2
Drug: Nintedanib — Continuous high dose
  Arms: Level 3

SUMMARY:
Phase I study. To determine the MTD (Maximum Tolerated Dose) of nintedanib + weekly Docetaxel in patients with locally advanced or metastatic lung adenocarcinoma after failure of platinum-based first line chemotherapy.

ELIGIBILITY:
Inclusion criteria:

-Patients with histologically/ cytologically confirmed locally advanced (Stage IIIB) or metastatic (Stage IV) lung adeno carcinoma after failure of first line platinum - based chemotherapy (patients with non-target lesion only are eligible).

First line chemotherapy may include continuation or switch maintenance therapy. One prior adjuvant and/or neoadjuvant chemotherapy line is accepted. Prior immunotherapy is allowed.

* ECOG inferior or equal to 1 at screening.
* Further inclusion criteria apply

Exclusion criteria:

* Patients who have received more than one prior line of chemotherapy (i.e. second or third line chemotherapy) for advanced or metastatic NSCLC.
* Patients known to be positive for activating Epidermal Growth Factor Receptor (EGFR) mutation or patients known to be positive for ALK translocation
* Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-03-07 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (4):
- France (2):
  - HOP d'Angers, Angers
  - HOP Jean Minjoz, Besançon
- Germany (2):
  - Pneumologisches Forschungsinstitut an der LungenClinic Grosshansdorf GmbH, Großhansdorf
  - Krankenhaus Martha-Maria Halle-Dölau gGmbH, Halle

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study is an open-label Phase I of oral nintedanib plus weekly docetaxel therapy in subjects with locally advanced or metastatic lung adenocarcinoma after failure of platinum-based first-line chemotherapy.
Pre-assignment Details: All subjects who signed informed consent were screened for eligibility prior to participation in the trial. Subjects were assigned to trial drug if they met all inclusion criteria and none of the exclusion criteria. Subjects attended a specialist site in oncology.
Groups:
- 150 mg Nintedanib + Docetaxel: In a treatment cycle of 28 days, 150 milligram (mg) nintedanib was administered orally twice a day with a dose interval of 12 hours with 250 milliliter (mL) of water after food intake except on the days of docetaxel infusion. Docetaxel (35 mg per square meter of body surface (mg/m2)) was administrated as a intravenous infusion over 60 minutes on Days 1, 8 and 15. The 28-day treatment cycles could be repeated until disease progression. In case of nintedanib-related adverse events, the dose of nintedanib was to be reduced to 100 mg twice a day, a second dose reduction was not allowed.
- 200 mg Nintedanib + Docetaxel: In a treatment cycle of 28 days, 200 milligram (mg) nintedanib was administered orally twice a day with a dose interval of 12 hours with 250 milliliter (mL) of water after food intake except on the days of docetaxel infusion. Docetaxel (35 mg per square meter of body surface (mg/m2)) was administrated as a intravenous infusion over 60 minutes on Days 1, 8 and 15. The 28-day treatment cycles could be repeated until disease progression. In case of nintedanib-related adverse events, the dose of nintedanib was to be reduced to 150 mg twice a day with a possible second dose reduction to 100 mg twice a day.
Period: Overall Study
Arm/Group | 150 mg Nintedanib + Docetaxel | 200 mg Nintedanib + Docetaxel
Started | 7 | 7
Completed | 0 | 1
Not Completed | 7 | 6
Not completed — Progressive disease | 6 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal from the trial | 0 | 1
Not completed — Lack of benefit and side effects | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): all subjects who received at least one dose of study medication. The TS was used for all safety and efficacy analyses
Groups:
- Total: Total of all reporting groups
Arm/Group | 150 mg Nintedanib + Docetaxel | 200 mg Nintedanib + Docetaxel | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (7.6) | 60.3 (7.8) | 63.6 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 5 | 5 | 10
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 5 | 5 | 10
  Not reported due to local law restrictions | 2 | 2 | 4
Race/Ethnicity, Customized [Number; unit: Participants]
  Not Hispanic or Latino | 5 | 5 | 10
  Not reported due to local law restrictions | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Nintedanib Administered in Combination With Docetaxel
Description: Maximum tolerated dose (MTD) of nintedanib administered in combination with docetaxel. The MTD was defined as the highest dose combination studied for which the incidence of DLTs was no more than 1 out of 6 subjects experiencing a DLT during the first treatment cycle i.e. the incidence of DLTs was no more than 17%. In case dose escalation reached dose level 3 (200 mg bid nintedanib administered without interruption on days of docetaxel infusion) and no more than 1 out of 6 subjects experienced a DLT during the first 28-day cycle at this dose level, dose level 3 was considered the MTD.
Time Frame: First treatment cycle, the first 28 days following the start of trial medication.
Population: Maximum tolerated dose (MTD) Evaluation Set: All subjects who received at least one dose of study medication and were evaluable for MTD determination.
Measure: Number; unit: milligram
Groups:
- Nintedanib + Docetaxel: Comprises all dose cohorts during the dose escalation phase. In a treatment cycle of 28 days, 150 milligram (mg) nintedanib was taken orally twice a day with a dose interval of 12 hours with 250 milliliter (mL) of water after food intake except on the days of docetaxel infusion. Docetaxel (35 mg per square meter of body surface (mg/m2)) was administrated as a intravenous infusion over 60 minutes on Days 1, 8 and 15. The 28-day treatment cycles could be repeated until disease progression.
Arm/Group | Nintedanib + Docetaxel
Number analyzed (Participants) | 12
milligram | NA — Maximum tolerated dose was not reached as recruitment of participants into the dose escalation part was not fully completed due to premature discontinuation of the study.

2. Primary Outcome: Number of Participants With Dose-limiting Toxicity (DLT) During the First Treatment Cycle
Description: Number of participants with DLT occurring during the first treatment cycle. DLT was defined as any of the following adverse events related to nintedanib:
  * Non-haematological drug-related Common Terminology Criteria for AEs (CTCAE) grade 3 or greater
  * diarrhoea CTCAE grade 2 for >7 days despite supportive care
  * nausea CTCAE grade 3 or greater despite supportive care
  * vomiting CTCAE grade 2 or greater despite supportive care
  * increase in Alanine aminotransferase (ALT) and/or Aspartate aminotransferase (AST) to CTCAE grade 3 or greater
  * A increase in ALT and/or AST to CTCAE grade 2 or greater in conjunction with
  * total bilirubin increase of CTCAE grade 1 or greater
  * Platelets <50 000/mm3 with bleeding (CTCAE ≥3)
  * neutropenia of any grade or duration accompanied by fever >38.5°C
  * neutropenia grade 4 without fever of >7 days duration
  * Inability to resume nintedanib dosing within 21 days after stopping due to toxicity.
Time Frame: First treatment cycle, the first 28 days following the start of trial medication.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg Nintedanib + Docetaxel | 200 mg Nintedanib + Docetaxel
Number analyzed (Participants) | 6 | 6
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: From first administration of study drug till the last administration + a residual effect period (REP) of 28 days, up to 330 days.
Description: Treated set (TS): all subjects who received at least one dose of study medication. The TS was used for all safety and efficacy analyses.
Arm/Group | 150 mg Nintedanib + Docetaxel | 200 mg Nintedanib + Docetaxel
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 3/7 | 2/7
Other Adverse Events (participants affected / at risk) | 6/7 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 150 mg Nintedanib + Docetaxel (N=7) | 200 mg Nintedanib + Docetaxel (N=7)
Nausea (Gastrointestinal disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Empyema (Infections and infestations) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 150 mg Nintedanib + Docetaxel (N=7) | 200 mg Nintedanib + Docetaxel (N=7)
Anaemia (Blood and lymphatic system disorders) | 3 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Lacrimation increased (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Abdominal rigidity (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 2 | 0
Condition aggravated (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 2
Mucosal inflammation (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 2 | 1
Pyrexia (General disorders) | 1 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Nail infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Transaminases increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Taste disorder (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 2 | 0
Onychalgia (Skin and subcutaneous tissue disorders) | 1 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Capillary leak syndrome (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Recruitment was prematurely discontinued after dose level 2 (200 milligram) due to difficulties in recruiting subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2015-11-04): https://cdn.clinicaltrials.gov/large-docs/93/NCT02668393/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-21): https://cdn.clinicaltrials.gov/large-docs/93/NCT02668393/SAP_001.pdf